CLINICAL TRIAL: NCT02696746
Title: Painful Channelopathies Study
Acronym: PCS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: University of Oxford (Other); Neuroscience Technologies S.L.P (Industry)
Responsible Party: Sponsor
Other Study IDs: 12/LO/0017
Record Dates: First submitted 2016-02-05; First posted 2016-03-02 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-02

CONDITIONS: Erythromelalgia; Pain Insensitivity, Congenital; Hereditary Sensory and Autonomic Neuropathies; Chronic Pain
MeSH Terms: conditions — Erythromelalgia; Pain Insensitivity, Congenital; Hereditary Sensory and Autonomic Neuropathies; Chronic Pain | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 1. The investigators will collect blood samples (30mls) from each subject, which will be stored at -800C in a locked freezer. They will sequence known genes associated with painful channelopathies: SCN9a and TRPA1. They will store DNA in order that it is possible that other candidate genes associated with pain can be tested.
  2. 3mm skin punch biopsies performed 10 cm above lateral malleolus for 2 different purposes:
     * Nerve fibre density measurement
     * Fibroblasts cultures as these represent a useful tool in the future as a source of cells the phenotype of which can be modulated for instance to generate induced pluripotent stem cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pain related conditions: Subjects with painful or painless conditions (observational study, no interventions)
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — No intervention

SUMMARY:
To understand the pathophysiological basis of heritable pain syndromes. This will consist of a number of components:

* Determine the genetic basis for heritable pain syndromes.
* Investigate the pain symptoms, psychological co-morbidity and quality of life in patients with heritable pain syndromes.
* Use quantitative sensory testing to investigate abnormalities in sensory processing.
* Use imaging modalities to investigate the neural correlates of pain perception in heritable channelopathies.
* In select patients to perform skin biopsy to determine if there has been any damage to C-fibres.
* To perform skin biopsy in order to culture fibroblasts and neural crest stem cells for future studies into the molecular basis of altered pain perception.
* To use neurophysiological tests, the axon reflex, and conditioning challenges to determine how peripheral nerves, in heritable channelopathies and unusual pain syndromes, have been altered.
* Microneurographic recordings for directly detecting the function of pain fibres in peripheral nerves. Knowledge gained from the study will be used to aid the further development of genetic testing and specific pain questionnaires for the diagnosis of heritable pain syndromes secondary to channelopathies.
* Ultimately better knowledge of underlying pathophysiology in these heritable pain conditions may inform the development of novel treatments.

DETAILED DESCRIPTION:
Very little is currently known about the sensory characteristics and central processing of pain in patients with heritable channelopathies. The investigators will carefully study the phenotype of such patients in terms of pain symptomatology, sensory processing as revealed by quantitative sensory testing and correlate this with genotype. In select patients the investigators will perform skin biopsy to determine whether there is any evidence of damage to small fibres and would also like to generate fibroblast and neural crest stem cell cultures for future studies of the molecular basis for channel dysfunction.

The study will provide new insights into the peripheral and central nervous system mechanisms involved in the processing of pain.

The investigators will restrict themselves to channelopathies causing somatic pain syndromes and will not be investigating migraine. The following conditions will be considered: Erythromelalgia, Paroxysmal extreme pain disorder, Familial episodic pain syndrome, patients with episodic pain symptoms for which a cause cannot be found and patients with reduced pain sensibility.

1.2.1 Quantitative sensory testing (QST)

QST is a method for accurately determining sensory thresholds in human skin and is particularly useful for determining dysfunction in the nociceptive smaller diameter nerve fibres, although the precise utility of QST in routine clinical neuropathic pain management perhaps requires some further evaluation. There is also increasing interest in using QST in combination with assessment of pain descriptors to give insights into the underlying pathophysiological mechanisms of chronic pain. For example, the presence of brush evoked dynamic allodynia indicates sensitisation at the spinal level. The investigators will use a standardized protocol developed by the german neuropathic pain consortium in which they have great experience. Only limited studies have been performed on inherited painful channelopathies in assessing sensory function. The investigators will correlate findings in QST with pain symptoms and quality of life. The investigators would like to see if specific abnormalities of sensory processing are associated with particular channelopathies.

1.2.2 Skin biopsy.

Measurement of intra epidermal nerve fibre density (IENFD) is a relatively simple assay which can be performed in relatively innocuous 3mm punch biopsies of skin, a routine dermatological investigation. Its utility in the assessment of small fibre function in peripheral neuropathies is clear. Peripheral neuropathies of diverse aetiologies are associated with reduced epidermal innervation density. The investigators have extensive experience in this technique which has minimal morbidity and would like to establish in painful channelopathies whether the anatomy of C-fibres innervating the skin is normal. Patients can opt out of this and still be included in the study. Fibroblasts can be cultured from 4mm skin biopsy (obtained as described above). These represent a useful tool in the future as a source of cells the phenotype of which can be modulated for instance to generate induced pluripotent stem cells followed by induction of neural crest differentiation in order to understand the molecular basis of altered pain perception. A further approach is to isolate neural crest stem cells directly from hair follicles a technique pioneered by Prof Sieber-Blum at Newcastle University. The investigators subsequently aim to generate sensory neurons from these cells and compare the behaviour of sensory neurons from control subjects to those generated from patients with heritable pain syndromes.

1.2.3 Electrodiagnostic tests

Electrodiagnostic tests: These assess the integrity of the peripheral large nerve fibres. Nerve conduction studies (NCS) are used extensively in clinical practice to diagnose peripheral neuropathies and are safe procedures in which the integrity of the axon and its myelin sheath are tested using external electrical stimuli. Threshold tracking techniques, the electrical threshold at which nerve respond to electrical stimulation, will also be used to study the peripheral nerves.

If NCS have been performed as part of the patient's routine medical care these results will be recorded.

Microneurography: Traditional nerve conduction studies only detect activity in the largest nerve fibres. To record from the smallest nerve fibres the investigators may perform microneurography. This is a minimally invasive technique in which the activity of single nerve fibre is recorded from peripheral nerves and is for directly detecting the function of pain fibres in peripheral nerves in humans. In this test a thin micro-electrode is placed next to the nerve fibres. This provides the only direct means to directly record C-fibre activity in humans. J Serra a co-investigator in this study and has a long track record in using microneurography.

1.2.4 Chemical challenges to measure the axon reflex and condition the sensory nervous system

As a further means of assessing the physiological integrity of the peripheral C fibers in patients suffering from unusual pain syndromes or reduced pain sensitivity the investigators will elicit an axon reflex. This reflex involves the transcutaneous application of agents such as histamine via iontophoresis. The histamine will stimulate the peripheral nerve endings of the small diameter C fibres. Their stimulation induces a vasodilatation, which is visible as a flare response of the skin. The evaluation of the extent of the flare response is used as an indication of the integrity of the small diameter C fibre population. If the subject has any allergies they will be excluded from this test.

Conditioning challenges are interventions that sensitise the peripheral nociceptive system in such a way that the nociceptive system either responds more vigorously to noxious stimuli (hyperalgesia) or responds to non-noxious stimuli (allodynia). The manner in which that peripheral nociceptive system responds provides important information as to the physiological functioning of the peripheral nociceptor system. The investigators will apply established conditioning challenges to the subjects' skin. Topical application of capsaicin and mustard oil are all well validated, established and safe conditioning challenges that sensitise peripheral nociceptors. Prof. David Bennett's group has extensive experience in using both conditioning challenges. In the only study to date investigating alteration of peripheral fibres after a conditioning challenge in heritable pain syndromes, mustard oil caused an increased area of hyperalgesia in individuals with Familial Episodic Pain Syndrome as compared to unaffected individuals. Applying these stimuli could lead to minor skin irritation and that is they will not be used if there is a history of skin allergy/sensitivity. In practice having performed such tests hundreds of times this has not been a problem.

1.2.5 Imaging the Human Brain in Pain

The advent of functional imaging techniques allowed researchers to begin to look within the human brain to observe what pain looks like in the brain. Initially, pain imaging research determined that pain is not processed by a single brain region but instead engages several distributed cortical areas. The group of brain regions that are most active during pain are commonly referred to as the 'pain matrix'. This includes: primary and secondary somatosensory cortices (SI, SII), insular, anterior cingulate, and prefrontal cortices and the thalamus.

However, pain is not purely a sensory event but is also reflective of how the person feels about their pain. Factors that vary widely across a population such as memories, emotion, pathology, genetics, and cognitive factors all directly affect how an individual experiences pain. In addition, the way a person responds to pain is modified heavily by what is appropriate for the situation. For example, a person in pain may hide how unpleasant the sensation is if they are uncomfortable in their surroundings. Because of this, the pain matrix provides an incomplete picture of what is happening in the brain during pain. Pain imaging studies have begun to validate this perspective. For example, Derbyshire and collaborators showed activation of the key pain matrix regions even when subjects were not in pain. From a study looking at chronic pain sufferers, it was shown that a series of other key brain regions were active that were outside the pain matrix. It is essential for brain imaging research to update the notion of the 'pain matrix' to account for these inconsistencies.

1.2.6 Psychological co-morbidity, quality of life and pain

Whilst some studies have examined aspects of pain in the context of nerve injury (and very rarely in relation to inherited channelopathies), these do not go beyond more than simple measurement of pain intensity or sensory characteristics and there is only a limited literature which has explored the interactions between pain, psychological status and quality of life. Neuropathic pain in general is associated with multiple psychological problems which impact upon quality of life. These include circadian rhythm disturbances (e.g. sleeping difficulty: moderate to severe in 60% of patients), lack of energy (55%), drowsiness (39 %) and difficulty in concentration (36%); similar findings have been specifically documented in erythromelalgia. A poor health perception, poor physical functioning, a high prevalence of role limitation (physical and emotional), as well as, depressive symptoms (based on the pain catastrophising scale and on the Center for Epidemiologic Studies Depression Scale) were all found in patients with Erythromelalgia. In general, beliefs and fears concerning the pain and its implications contribute substantially to determining mood and behaviour. Since neuropathic pain is relatively common in the context of peripheral neuropathy the question arises as to what extent pain is the driver of these co-morbidities - the answer to this is not known, but large randomised controlled trials of analgesic interventions in neuropathic pain states indicate that as pain intensity reduces so does the severity of these co-morbidities. To answer this question the investigators will first need to identify specific tools for the measurement of neuropathic pain co-morbidity in the context of painful channelopathies this is one of the aims of this proposal and they will evaluate a variety of existing assessment tools. Another issue is that it is likely that psychological co-morbidity influences the self reporting of pain intensity, which is a usual primary outcome measure in clinical trials of neuropathic pain analgesic agents.

The investigators will use a battery of psychological instruments to determine the psychological and quality of life in those subjects with painful channelopathies.

1.2.7 Blood samples

The investigators will collect blood samples (30mls) from each subject, which will be stored at -80 degrees Celsius in a locked freezer. They will sequence known genes associated with painful channelopathies: SCN9a and TRPA1. The investigators will store DNA in order that it is possible that other candidate genes associated with pain can be tested.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are ≥16 years of age who have a set of symptoms that resemble those seen on Paroxysmal Extreme Pain Disorder, Familial Episodic Pain Syndrome or Erythromelalgia.
* Patients already with the diagnosis of Paroxysmal Extreme Pain Disorder or Familial Episodic Pain Syndrome or Erythromelalgia.
* Patients with reduced pain sensibility.
* First degree relatives of patients who meet diagnostic criteria for Paroxysmal Extreme Pain Disorder, Familial Episodic Pain Syndrome, Erythromelalgia or inability to experience pain.
* Patients who do not fulfill any of the exclusion criteria.

Exclusion Criteria:

* Pregnant subjects.
* Subjects with insufficient command of English to obtain consent from or to complete the study questionnaires.
* Subjects with insufficient mental capacity to obtain consent from or to complete the study questionnaires.
* Subjects with concurrent severe psychological or psychiatric disorders, specially those patients with severe claustrophobia.
* Patients with moderate to severe pain arising as a consequence of other disorders causing pain but that are not associated with those mentioned before as channelopathies.
* Patients with central nervous system diseased that may complicate the somatosensory testing.
* The skin biopsy procedure, will not be conducted on those patients with contraindications to do so i.e. anticoagulation therapy, skin infections, etc; that might result in adverse outcomes (if the subject decides to decline the skin biopsy, the inclusion on the study will not be affected).
* The functional magnetic resonance imaging (fMRI) component will not be performed in subjects that had medical interventions with any device likely to be damaged or moved from its place, at any moment during the fMRI scanning procedure (including cerebral coils or clips, heart pacemakers or defibrillators, heart valve prosthesis, medicine infusion pumps, inner ear implants, neural stimulators, brain shunts, joint replacements/ large metal implants, stents in the heart or arteries, some implants, or some intra-uterine contraceptive devices.
* Those patients that in the concept of the research team unsuitable for participation in the study.
* For those undergoing microneurography presence of edema (swelling) or any skin condition at the ankle level that may interfere with the microneurography procedure.
* Patients with a history of skin allergy or sensitivity will not undergo testing of axon reflex or conditioning challenges.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and family members affected by chanelopathic pain related conditions.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-02; Primary Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Pain score | Day 7
  Seven days pain diary of 4 or above. Patients will have 7-days pain diaries with a numeric rating scale from 0 to 10.

SECONDARY OUTCOMES:
Age | Day 1
  Number of years
Gender | Day 1
  Chromosome gender (male/female)
Ethnicity | Day 1
  Ethnic group
Detailed medical history | Day 1
  Number and name of medications that were taken previously by the patient
Pain related anxiety | Day 1
  Patients will answer the Pain Anxiety Symptoms Scale (PASS-20)
Measures of quality of life | Day 1
  Patients will answer the 36-Item Short Form Survey -quality of life questionnaire-
Measures of sleep interference | Day 1
  Sleep quality is assessed through the use of questionnaires
Nerve Conduction Studies | Day 1
  Neurophysiology will be conducted to assess nerve integrity. Amplitude will be measured in microvolts.
Nerve Conduction Studies | Day 1
  Neurophysiology will be conducted to assess nerve integrity. Latency will be measured in milliseconds.
Microneurography Studies | Day 1
  This is a minimally invasive technique in which the activity of single nerve fibre is recorded from peripheral nerves and is for directly detecting the function of pain fibres in peripheral nerves in humans.
Sensory Thermal Thresholds | Day 1
  Thermal thresholds will be measured in degrees centigrade
Sensory Mechanical Detection Thresholds | Day 1
  Mechanical Detection Thresholds will be measured in millinewtons
Intra-Epidermal Nerve Fibre density | Day 1
  Measurement of nerve fibres in the skin of patients (taken depending of the pain related area)
Skin biopsy | Day 1
  Collection and culture of fibroblasts and neural crest stem cells for assessing differences in the rheobase measured in amperes.
Axon reflex measurement | Day 1
  Application of agents such as histamine via iontophoresis which will stimulate the peripheral nerve endings of C fibres inducing a vasodilatation, which is visible as a flare response of the skin (area in square centimeters with flare).
Functional Magnetic Resonance Imaging | Day 30
  Brain activity related to the pain condition
Blood samples - DNA | Within 6 months of visit
  Blood samples coupled with detailed phenotype data will investigate potential gene associations in the development of painful or painless conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuffield Department of Clinical Neurosciences, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Result] Ramirez JD, Habib AM, Cox JJ, Themistocleous AC, McMahon SB, Wood JN, Bennett DL. Null mutation in SCN9A in which noxious stimuli can be detected in the absence of pain. Neurology. 2014 Oct 21;83(17):1577-80. doi: 10.1212/WNL.0000000000000913. Epub 2014 Sep 24. No abstract available. PMID 25253744